CLINICAL TRIAL: NCT03292796
Title: A Randomised Control Study to Investigate if the Continuation of Prostaglandin Analogue Treatments in the Post-operative Phase of Glaucoma Patients Undergoing Cataract Surgery Increases the Incidence of Cystoid Macular Oedema.
Brief Title: RCT to Investigate if Prostaglandin Analogue Drops Increase the Risk of Cystoid Macular Oedema After Cataract Surgery.
Acronym: CMO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Julie Dawson (Other)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014OPH03L(104-0614); REC 15/EE/0239 (Other: Research Ethics Committee)
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Open Angle Glaucoma and Cataract
Keywords: Open Angle Glaucoma; Cataract; Phacoemulsification,; Cystoid Macular Oedema,; Prostaglandin Analogues
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract; Macular Edema | interventions — Prostaglandins

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Who Masked: Outcomes Assessor
Masking Description: * The patient is not masked as to treatment group and are aware of whether they are to continue or stop the PGA drops
  * The care providers are not masked as to treatment group
  * Outcome assessors are masked as to the patient's treatment group for their analysis of the OCT scans over the 4 week peri-operative period.
    * The scans are recorded with only the randomised identifier.
    * This is to reduce bias in the analysis of the scans
    * Unmasking of each patient will occur after their analysis of their week 4 OCT scan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stop prostaglandin eye drops post op (Other): Stop prostaglandin eye drops post operatively. Prostaglandins either stopped or continued after cataract surgery. Latanoprost Travaprost Bimatoprost Tafluprost
  Interventions: Drug: Prostaglandins
- Continue prostaglandin eye drops post op (Other): Continue prostaglandin eye drops post operatively Prostaglandins either stopped or continued after cataract surgery. Latanoprost Travaprost Bimatoprost Tafluprost
  Interventions: Drug: Prostaglandins

INTERVENTIONS:
Drug: Prostaglandins
  Other Names: Latanoprost Travaprost Bimatoprost Tafluprost

SUMMARY:
Post-operative cystoid macular oedema (CMO) is a common complication causing visual loss following routine cataract surgery. This complication is more prevalent in eyes with excessive inflammation as they heal from surgery.

Prostaglandin analogues (PGA) are the commonest first line drugs used in the long-term treatment of primary open angle glaucoma (POAG)- where they reduce the pathologically high pressure in the eye. Prostaglandins are inflammatory mediators.

In the post-operative care of glaucoma patients undergoing cataract surgery, there is a clinical dilemma whether to stop or continue the use of prostaglandin eye drops. Clinical practice is completely dichotomized between continuing and stopping PGA treatment in the postoperative period. There is conflicting scientific literature on the effect of PGA on the incidence of CMO; and only a single randomized control trial (Miyake K, Arch Ophthalmol 1999, 117:34-40), where the post operative regime is not applicable to present practice, compared the incidence of CMO following routine cataract surgery in POAG on PGA.

DETAILED DESCRIPTION:
This study aims to answer the common clinical question of whether or not to stop PGA after routine cataract surgery. Cataract surgery is the commonest operation performed on the NHS and the prevalence of glaucoma is 5% in the population over 80 years old. Thus the clinical dilemma is a common one.

A current literature search reveals that a divided opinion over whether PGAs do increase the incidence of CMO. No study has yet established a causal relationship between the use of PGAs and the development of CMO. Anecdotal reports and small case series have associated peri-operative PGA use with the occurrence of CMO (Henderson BA et al, 2007 J Cataract Refract Surg 33:1550-1558; Moroi SE et al, 1999, Ophthalmology 106:1024-1029). Whilst, in direct contrast, other authors argue CMO as a rare phenomenon and the causative relationship is debated (Schumer RA et al 2000, Curr Opin Ophthalmol 11:94-100; Miyake K et al 2003 J Cataract Refract Surg 29:1800-1810)

The most similar previous study to the one proposed, was by Miyake K et al. (Arch Ophthalmol 1999, 117:34-40). The key difference, though, is in the postoperative drop regime of fluorometholone and diclofenac in that paper and current UK clinical practice of using dexamethasone. In terms of study design, this paper used an invasive method of investigating CMO by fundus fluorescein angiography compared to OCT proposed here.

A recent case report by Agange N & Mosaed S (Journal of Ophthalmology, 2010) concludes with 'conclusions about causal relationships cannot be made without well-designed, prospective clinical trials addressing this issue'.

This study will therefore use drops that are routinely used in current UK clinical practice and add to the body of evidence that helps answer the question should PGAs be continued after cataract surgery so as to prevent the progression of glaucoma in patients.

* Aim

  * This study investigates if the occurrence of CMO after cataract surgery is affected by the use of PGA drops by patients with glaucoma
  * The null hypothesis states there is no increase in the incidence of CMO on OCT scanning in the 4 weeks following cataract surgery whether PGA eye drops continue or are stopped.
* Design

  * Randomised control study with parallel group design
  * Single masking of outcome assessors

ELIGIBILITY:
Inclusion Criteria:

* Primary open-angle glaucoma and ocular hypertensive subjects undergoing cataract surgery (routine phacoemulsification and intraocular lens implantation) AND on current topical glaucoma treatment with a prostaglandin analogue eye drop for at least 2 months prior to cataract surgery.
* Subjects capable of giving informed consent

Exclusion Criteria:

* Subjects with additional risk factors for macula oedema (eg. diabetic retinopathy, previous macula oedema, uveitis)
* Subjects with advanced glaucoma

  * Advanced visual field loss (Humphrey Mean Deviation >-12dB)
  * Advanced glaucomatous disc changes (vertical cup-to-disc ratio >0.9)
* Subjects with non-controlled intraocular pressure (IOP) (pre-operative IOP >22 mmHg)
* Any contra-indication to the use of topical prostaglandin drops
* Any contra-indication to the use of routine post-operative dexamethasone 0.1% eye drops
* Pregnancy
* Patients unable to give informed consent
* Intra-operative complication during cataract phacoemulsification and intraocular lens implantation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
Occurrence of cystoid macula oedema (CMO) at 4 weeks post operatively | 4 weeks post operatively
  Occurrence of cystoid macula oedema (CMO) at 4 weeks post operatively.Cystoid macular oedema will be defined as an increase in the central macula thickness on the OCT with characteristic intraretinal changes in the 4 weeks following surgery.

SECONDARY OUTCOMES:
Intraocular pressure (IOP) at 4 weeks post-operatively. | 4 weeks post operatively
  Intraocular pressure (IOP) at 4 weeks post-operatively. Intraocular pressure will be measured by Goldmann applanation tonometry, the standard method used in clinical practice to monitor glaucoma. This forms part of the standard post-operative examination following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nuwan Niyadurupola, Consultant, Principal Investigator — Consultant Ophthalmologist
Locations (1):
- Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agange N, Mosaed S. Prostaglandin-induced cystoid macular edema following routine cataract extraction. J Ophthalmol. 2010;2010:690707. doi: 10.1155/2010/690707. Epub 2010 Nov 7. PMID 21076526
- [Background] Henderson BA, Kim JY, Ament CS, Ferrufino-Ponce ZK, Grabowska A, Cremers SL. Clinical pseudophakic cystoid macular edema. Risk factors for development and duration after treatment. J Cataract Refract Surg. 2007 Sep;33(9):1550-8. doi: 10.1016/j.jcrs.2007.05.013. PMID 17720069
- [Background] Miyake K, Ota I, Maekubo K, Ichihashi S, Miyake S. Latanoprost accelerates disruption of the blood-aqueous barrier and the incidence of angiographic cystoid macular edema in early postoperative pseudophakias. Arch Ophthalmol. 1999 Jan;117(1):34-40. doi: 10.1001/archopht.117.1.34. PMID 9930158
- [Background] Miyake K, Ibaraki N, Goto Y, Oogiya S, Ishigaki J, Ota I, Miyake S. ESCRS Binkhorst lecture 2002: Pseudophakic preservative maculopathy. J Cataract Refract Surg. 2003 Sep;29(9):1800-10. doi: 10.1016/s0886-3350(03)00560-1. PMID 14522305
- [Background] Moroi SE, Gottfredsdottir MS, Schteingart MT, Elner SG, Lee CM, Schertzer RM, Abrams GW, Johnson MW. Cystoid macular edema associated with latanoprost therapy in a case series of patients with glaucoma and ocular hypertension. Ophthalmology. 1999 May;106(5):1024-9. doi: 10.1016/S0161-6420(99)00528-X. PMID 10328408
- [Background] Schumer RA, Camras CB, Mandahl AK. Latanoprost and cystoid macular edema: is there a causal relation? Curr Opin Ophthalmol. 2000 Apr;11(2):94-100. doi: 10.1097/00055735-200004000-00005. PMID 10848227